CLINICAL TRIAL: NCT02896140
Title: The Effect of Dairy Product Consumption on Glycemic Control, Body Weight and Cardiovascular Risk Factors in Patients Enrolled in the Joslin Weight Achievement and Intensive Treatment (Why WAIT) Program: A Prospective Cohort Study
Brief Title: Effect of Dairy Consumption on Glycemic Control, Body Weight and Cardiovascular Risk Factors
Status: Completed | Type: Observational
Sponsor: Joslin Diabetes Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-07
Record Dates: First submitted 2016-04-26; First posted 2016-09-12 (Estimated); Last update posted 2019-03-01 (Actual); Status verified 2019-02

CONDITIONS: Diabetes Mellitus, Type 2; Obesity
Keywords: Type 2 diabetes; Obesity; Nutrition; Dairy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Type 2 diabetes in WhyWAIT Program: Patients with type 2 diabetes who are participating in Joslin Diabetes Center's 12-week intensive diabetes weight management program (WhyWAIT).
  Interventions: Other: Type 2 diabetes in WhyWAIT Program

INTERVENTIONS:
Other: Type 2 diabetes in WhyWAIT Program — The sum of servings per day of milk, cheese, yogurt, and other dairy foods.

SUMMARY:
The aim of this study is to determine the relationship between the percentage of calories from dairy intake and long-term glycemic control and weight maintenance in patients with type 2 diabetes who participate in an intensive lifestyle intervention program.

The investigators hypothesize that overweight and obese patients with type 2 diabetes who consume higher percentage of calories from dairy products during intensive lifestyle intervention programs have better glycemic control and maintenance of weight loss as compared to those who consume lower percentage of calories from dairy products.

DETAILED DESCRIPTION:
This is a prospective, observational clinical study where the daily intake of dairy products will be recorded and analyzed in 50 overweight/obese subjects with type 2 diabetes enrolled in the Weight Achievement and Intensive Treatment (Why WAIT) program. The Weight Achievement and Intensive Treatment (Why WAIT) program is a 12-week multidisciplinary program developed by Joslin Diabetes Center for intensive diabetes weight management in clinical practice. It includes the following components that are provided in a group setting: (1) intensive medical treatment provided by an endocrinologist and a registered nurse; (2) a structured dietary plan provided by a registered dietitian; (3) an individualized exercise training program provided by an exercise physiologist; (4) cognitive behavioral modification provided by a behavioral therapist.

Participants will be enrolled in this study for a period of 24 weeks. They will attend the Weight Achievement and Intensive Treatment (Why WAIT) program during the first 12 weeks of the study and will be followed for another 12 weeks after the program (the maintenance phase). During the intervention phase, participants will receive group education on a weekly basis for 12 consecutive weeks. During maintenance phase, participants will receive a monthly, 15 minute long, follow up phone call from the study dietitian.

Participants will be instructed to complete a 3-day food log before each visit. They will also be asked to record their dairy intake on a daily basis in a dedicated log book. These logs will be collected and analyzed by the study dietitian. Dairy consumption will be calculated as the sum of servings per day of milk, cheese, yogurt, and other dairy foods.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is participating in the Weight Achievement and Intensive Treatment (Why WAIT) program
2. Subject is male or female ages 18-75
3. Subject has type 2 diabetes for at least three months prior to screening and treated with any antihyperglycemic medication

Exclusion Criteria:

1. Subject is pregnant or lactating
2. Subject has a heart pacemaker

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in Joslin Diabetes Center's Weight Achievement and Intensive Treatment (Why WAIT) program
Sampling Method: Probability Sample
Enrollment: 51 (Actual)
Dates: Start 2016-04; Primary Completion 2018-07 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1C (A1C) | 24 weeks

SECONDARY OUTCOMES:
Change in body weight | 24 weeks
Change in low-density lipoprotein (LDL) | 24 weeks
Change in high-density lipoprotein (HDL) | 24 weeks
Change in total cholesterol | 24 weeks
Change in triglycerides | 24 weeks
Change in fasting plasma glucose | 24 weeks
Change in Homeostatic model assessment (HOMA) insulin resistance (IR) index | 24 weeks
Height in meters | 24 weeks
Change in body fat percentage | 24 weeks
Change in fat free mass | 24 weeks
Change in total body water | 24 weeks
Change in waist circumference | 24 weeks
Change in trunk fat percentage | 24 weeks
Change in visceral fat level | 24 weeks
Change in blood pressure | 24 weeks
Change in c-reactive protein level | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Osama Hamdy, MD, PhD, Principal Investigator — Joslin Diabetes Center
Locations (1):
- Joslin Diabetes Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided